CLINICAL TRIAL: NCT00666302
Title: A Randomized, Investigator Blinded Study of Protopic (Tacrolimus) Ointment Vs. Elidel (Pimecrolimus) Cream in Patients With Atopic Dermatitis
Brief Title: A Comparison Study Between Protopic (Tacrolimus) Ointment and Elidel (Pimecrolimus) Cream in Treating Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-02-004
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; Protopic; Elidel
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus; pimecrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment
- 2 (Active Comparator)
  Interventions: Drug: pimecrolimus cream

INTERVENTIONS:
Drug: tacrolimus ointment — topical
  Other Names: Protopic; FK506 ointment
  Arms: 1
Drug: pimecrolimus cream — topical
  Other Names: Elidel
  Arms: 2

SUMMARY:
A study to compare efficacy of Protopic Ointment to that of Elidel Cream in treating patients with Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Atopic Dermatitis rated at least mild using the Investigator's Global Atopic Dermatitis Assessment involving a minimum of 5% of the body surface area
* Negative pregnancy test and agrees to practice effective birth control during the study

Exclusion Criteria:

* Skin disorder other than Atopic Dermatitis in the areas to be treated
* Extensive scarring or pigmented lesions in the areas to be treated that would interfere with rating of efficacy parameters
* Clinically infected Atopic Dermatitis at baseline
* Likely to require systemic corticosteroids; or likely to require intranasal or inhaled corticosteroids for an off-label indication or at higher doses than the maximum labeled dosing for the drug
* Known hypersensitivity to macrolides or any excipient of either study medication
* Chronic condition which is either not stable or not well controlled
* Pregnant or breast feeding an infant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2002-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) | 6 Weeks

SECONDARY OUTCOMES:
Investigator's Global Atopic Dermatitis Assessment (IGADA) | 6 Weeks
Patient's evaluation of itch | 6 Weeks
Body surface area affected | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Director — Astellas Pharma US, Inc.
Locations (14):
- United States (13):
  - Birmingham, Alabama
  - San Francisco, California
  - Kansas City, Kansas
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - New York, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Kirsner RS, Heffernan MP, Antaya R. Safety and efficacy of tacrolimus ointment versus pimecrolimus cream in the treatment of patients with atopic dermatitis previously treated with corticosteroids. Acta Derm Venereol. 2010;90(1):58-64. doi: 10.2340/00015555-0748. PMID 20107727
- [Background] Paller AS, Lebwohl M, Fleischer AB Jr, Antaya R, Langley RG, Kirsner RS, Blum RR, Rico MJ, Jaracz E, Crowe A, Linowski GJ; US/Canada Tacrolimus Ointment Study Group. Tacrolimus ointment is more effective than pimecrolimus cream with a similar safety profile in the treatment of atopic dermatitis: results from 3 randomized, comparative studies. J Am Acad Dermatol. 2005 May;52(5):810-22. doi: 10.1016/j.jaad.2004.12.038. PMID 15858471
- [Background] Fleischer AB Jr, Abramovits W, Breneman D, Jaracz E; US/Canada tacrolimus ointment study group. Tacrolimus ointment is more effective than pimecrolimus cream in adult patients with moderate to very severe atopic dermatitis. J Dermatolog Treat. 2007;18(3):151-7. doi: 10.1080/09546630701287332. PMID 17538803